CLINICAL TRIAL: NCT00545402
Title: A Randomized, Open Label Study Comparing the Effect of CellCept With Therapeutic Drug Monitoring, Tacrolimus and a Corticosteroid-sparing Regimen Versus Fixed Dose CellCept, Tacrolimus and Corticosteroids Maintained up to 6 Months, on Acute Rejection and Safety in Liver Transplant Patients.
Brief Title: A Study of CellCept (Mycophenolate Mofetil) in Combination Therapy in Liver Transplant Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21273
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-06

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Mycophenolic Acid; Tacrolimus; Adrenal Cortex Hormones; Methylprednisolone Hemisuccinate; Prednisone

ARMS (2):
- MMF, Adjusted Dose; Tacrolimus; Corticosteroids (Experimental): Participants received mycophenolate mofetil (MMF) 3 grams per day (g/d), orally (PO), twice per day (BID) with meals from Day 0 to Day 4; the dose was adjusted based on total exposure (AUC) using the Bayesian method with limited sampling strategy on Days 5 and 14, Months 1, 13, 6, 9, and 12. Participants also received tacrolimus adjusted to a target trough level of 8 to (-) 12 nanograms per milliliter (ng/mL) from Day 0 to Month 1; the dose was adjusted to reach a target trough level of 3-8 ng/mL from the end of Month 1 through Month 12. Participants also received corticosteroids 10-15 milligrams per kilogram (mg/kg), intravenously (IV), pre-operation on Day 0.
  Interventions: Drug: Mycophenolate mofetil, adjusted dose; Drug: Tacrolimus; Drug: Corticosteroids, IV
- MMF, Standard Dose; Tacrolimus; Corticosteroids (Active Comparator): Participants received MMF 2 g/d, PO, BID with meals from Day 0 to Month 12. Participants also received tacrolimus adjusted to a target trough level of 8-12 ng/mL from Day 0 to Month 1; the dose was reduced to reach a target trough level of 3-8 ng/mL from the end of Month 1 through Month 12. Participants also received corticosteroids 10-15 mg/kg, IV, pre-operation on Day 0; followed by 20 mg/d, PO, 4 times per day (QDS) from Day 0 through Month 1; 15 mg/d, PO, 3 times per day (TID) from the end of Month 1 through Month 2; 10 mg/d, PO, BID from the end of Month 2 through Month 3; and 5 mg/d once per day from the end of Month 3 through Month 6.
  Interventions: Drug: Tacrolimus; Drug: Corticosteroids, IV; Drug: Mycophenolate mofetil, Standard dose; Drug: Corticosteroids, PO

INTERVENTIONS:
Drug: Mycophenolate mofetil, adjusted dose — 3 g/d PO BID during meals from Day 0 to Day 4, followed by dose adjustment based on AUC using the Bayesian method with limited sampling strategy on Days 5 and 14, Months 1, 13, 6, 9, and 12.
  Other Names: CellCept
  Arms: MMF, Adjusted Dose; Tacrolimus; Corticosteroids
Drug: Tacrolimus — Target trough level of 8-2 ng/mL from Day 0 to Month 1, adjusted to a target trough level of 3-8 ng/mL from the end of Month 1 through Month 12
Drug: Corticosteroids, IV — 10-15 mg/kg IV pre-operation on Day 0
  Other Names: Solu-Medrol
Drug: Mycophenolate mofetil, Standard dose — 2 g/d PO BID during meals from Day 0 to Month 12
  Other Names: CellCept
  Arms: MMF, Standard Dose; Tacrolimus; Corticosteroids
Drug: Corticosteroids, PO — 20 mg/d QDS from Day 0 through Month 1; 15 mg/day, TID from the end of Month 1 through Month 2; 10 mg/d BID from the end of Month 2 through Month 3; and 5 mg/d once per day from the end of Month 3 through Month 6.
  Other Names: Cortancyl
  Arms: MMF, Standard Dose; Tacrolimus; Corticosteroids

SUMMARY:
This 2 arm study will compare the efficacy and safety of two CellCept-containing treatment regimens in de novo liver transplant patients. Patients will be randomized into one of two groups, to receive either CellCept (at a starting dose of 3g/day po, adjusted according to exposure) standard dose tacrolimus and corticosteroids (10-15 mg/kg i.v. on day 0), or fixed dose CellCept 2g/day po, standard dose tacrolimus and corticosteroids (10-15mg/kg i.v. on day 0, then reducing from 20mg to 5mg over 6 months, and discontinuing after 6 months). The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* recipient of a first orthotopic liver transplant.

Exclusion Criteria:

* history of organ transplants;
* patient receiving a multi-organ transplant;
* calculated creatinine clearance <=30mL/min before transplant;
* leukocyte count < 2000/mm3 at randomization;
* history of cancer within past 5 years, except for successfully treated basal cell or squamous cell cancer, or in situ cervical cancer;
* pregnant or breast-feeding females, or females of childbearing age not using effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- France (15):
  - Besançon
  - Bordeaux
  - Caen
  - Clichy
  - Créteil
  - Grenoble
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Nice
  - Paris
  - Rennes
  - Toulouse
  - Villejuif

RESULTS

PARTICIPANT FLOW:
Groups:
- Adjusted Mycophenolate Mofetil (MMF)+Tacrolimus+Corticosteroid: Participants received MMF tablets or capsules, 3 grams per day (g/d), orally (PO), twice daily (BID) with meals from Day 0 to Day 4; thereafter the dose was adjusted based on total exposure (area under the concentration-time curve [AUC]) using the Bayesian method with limited sampling strategy on Days 5 and 14 and Months 1, 3, 6, 9, and 12. Participants also received tacrolimus capsules, adjusted to a target trough level of 8-12 nanograms per milliliter (ng/mL) from Day 0 through Month 1; the dose was adjusted to reach a target trough level of 3-8 ng/mL from the end of Month 1 through Month 12. Participants also received an intravenous (IV) bolus of methylprednisolone 10-15 milligrams per kilogram (mg/kg) pre-operative on Day 0 per standard practice of the center.
- Fixed-Dose MMF + Tacrolimus + Corticosteroid (CS): Participants received MMF capsules or tablets, 2 g/d, PO, BID with meals from Day 0 to Month 12; tacrolimus capsules, adjusted to a target trough level of 8-12 ng/mL from Day 0 to Month 1; the dose was reduced to reach a target trough level of 3-8 ng/mL from the end of Month 1 through Month 12; and IV bolus of prednisone, 10-15 mg/kg, pre-operative on Day 0 followed by prednisone tablets, 20 mg/d, PO, from Day 0 through Month 1; 15 mg/d, PO, from the end of Month 1 through Month 2; 10 mg/d, PO, from the end of Month 2 through Month 3; and 5 mg/d from the end of Month 3 through Month 6. Prednisone was discontinued from Month 7 through end of treatment.
Period: Overall Study
Arm/Group | Adjusted Mycophenolate Mofetil (MMF)+Tacrolimus+Corticosteroid | Fixed-Dose MMF + Tacrolimus + Corticosteroid (CS)
Started | 90 | 90
Completed | 56 | 61
Not Completed | 34 | 29
Not completed — Discontinuation of treatment | 17 | 9
Not completed — Use of unauthorized immunosuppressant | 8 | 7
Not completed — Death | 5 | 7
Not completed — Graft loss | 2 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Reason not specified | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population includes all randomized participants who received at least 1 dose of MMF.
Groups:
- Adjusted MMF + Tacrolimus + CS: Participants received MMF tablets or capsules, 3 g/d, PO, BID with meals from Day 0 to Day 4; thereafter the dose was adjusted based on total exposure (AUC) using the Bayesian method with limited sampling strategy on Days 5 and 14 and Months 1, 3, 6, 9, and 12. Participants also received tacrolimus capsules, adjusted to a target trough level of 8-12 ng/mL from Day 0 through Month 1; the dose was adjusted to reach a target trough level of 3-8 ng/mL from the end of Month 1 through Month 12. Participants also received an IV bolus of methylprednisolone 10-15 mg/kg pre-operative on Day 0 per standard practice of the center.
- Fixed-Dose MMF + Tacrolimus + CS: Participants received MMF capsules or tablets, 2 g/d, PO, BID with meals from Day 0 to Month 12; tacrolimus capsules, adjusted to a target trough level of 8-12 ng/mL from Day 0 to Month 1; the dose was reduced to reach a target trough level of 3-8 ng/mL from the end of Month 1 through Month 12; and IV bolus of prednisone, 10-15 mg/kg, pre-operative on Day 0 followed by prednisone tablets, 20 mg/d, PO, from Day 0 through Month 1; 15 mg/d, PO, from the end of Month 1 through Month 2; 10 mg/d, PO, from the end of Month 2 through Month 3; and 5 mg/d from the end of Month 3 through Month 6. Prednisone was discontinued from Month 7 through end of treatment.
- Total: Total of all reporting groups
Arm/Group | Adjusted MMF + Tacrolimus + CS | Fixed-Dose MMF + Tacrolimus + CS | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (8.5) | 55.1 (8.3) | 54.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 74 | 71 | 145

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treated Biopsy Proven Acute Rejection (BPAR) According to Banff Criteria up to 12 Months Post-Transplant
Description: Banff criteria required at least 2 of the 3 following features for a histopathological diagnosis of acute rejection: portal inflammation, bile duct inflammation, and venous endothelial inflammation. Each item was graded from 0 to 3 where 0 equals (=) mild, 2 = moderate, and 3 = severe. The sum of the 3 individual scores, from 0 to 9, corresponded to the Rejection Activity Index (RAI). If RAI = 0, 1, or 2, there was no evidence of rejection. If RAI = 3, there was borderline acute rejection. If RAI = 4 or 5, there was mild acute rejection. If RAI = 6 or 7, there was moderate acute rejection. If RAI = 8 or 9, there was severe acute rejection.
Time Frame: Days 0, 5, and 14, Month 1, 2, 3, 6, 9, and 12, 28 days after Month 12 or last dose of study treatment, and 6 and 12 months after the last dose of study treatment
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Adjusted MMF + Tacrolimus + CS | Fixed-Dose MMF + Tacrolimus + CS
Number analyzed (Participants) | 87 | 87
percentage of participants | 8.0 | 8.2

2. Secondary Outcome: Percentage of Participants With Graft Loss
Description: Graft survival was defined as the time between the randomization date and the graft loss date. Participants were censored at the date of last follow up, the date of last contact or premature withdrawal, and date of death.
Time Frame: as for outcome 1
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Adjusted MMF + Tacrolimus + CS | Fixed-Dose MMF + Tacrolimus + CS
Number analyzed (Participants) | 90 | 90
percentage of participants | 2.2 | 5.6
Statistical Analysis 1: Comparison: Adjusted MMF + Tacrolimus + CS vs Fixed-Dose MMF + Tacrolimus + CS; Test type: Superiority or Other; p = 0.2611, Log Rank

3. Secondary Outcome: Graft Survival
Description: The median time, in months, between randomization and graft loss event. Participants were censored at the date of last follow up, the date of last contact or premature withdrawal, and date of death.
Time Frame: as for outcome 1
Population: ITT population
Measure: Median (Full Range); unit: months
Arm/Group | Adjusted MMF + Tacrolimus + CS | Fixed-Dose MMF + Tacrolimus + CS
Number analyzed (Participants) | 90 | 90
months | 12.9 [0.0 to 24.5] | 12.9 [0.0 to 20.2]

4. Secondary Outcome: Overall Survival (OS) at Month 12 - Percentage of Participants With an Event
Description: OS was defined as the time between the date of randomization and death up to Month 12. Participants were censored at the date of last follow up and the date of last contact or premature withdrawal.
Time Frame: Days 0, 5, and 14, Month 1, 2, 3, 6, 9, and 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Adjusted MMF + Tacrolimus + CS | Fixed-Dose MMF + Tacrolimus + CS
Number analyzed (Participants) | 90 | 90
percentage of participants | 8.9 | 11.1
Statistical Analysis 1: Comparison: Adjusted MMF + Tacrolimus + CS vs Fixed-Dose MMF + Tacrolimus + CS; Test type: Superiority or Other; p = 0.7091, Log Rank

5. Secondary Outcome: Overall Survival at Month 12
Description: The median time, in months, between randomization and OS event. Participants were censored at the date of last follow up and the date of last contact or premature withdrawal.
Time Frame: Days 0, 5, and 14, Month 1, 2, 3, 6, 9, and 12
Population: ITT population
Measure: Median (Full Range); unit: months
Arm/Group | Adjusted MMF + Tacrolimus + CS | Fixed-Dose MMF + Tacrolimus + CS
Number analyzed (Participants) | 90 | 90
months | 12.9 [0.0 to 24.5] | 12.9 [0.1 to 20.2]

6. Secondary Outcome: Percentage of Participants by Graft Histology at 12 Months Post-Transplant - Central Review
Description: The percentage of participants with biopsies of grafts evaluated by central review and scored according to Banff criteria at Month 12 post-transplant.
Time Frame: Days 0, 5, and 14, Month 1, 2, 3, 6, 9, and 12
Population: ITT population; only participants with evaluable biopsies were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Adjusted MMF + Tacrolimus + CS | Fixed-Dose MMF + Tacrolimus + CS
Number analyzed (Participants) | 42 | 35
percentage of participants
  Normal liver | 4.8 | 11.4
  Minor lesions | 4.8 | 17.1
  Acute rejection | 0.0 | 0.0
  Chronic rejection | 7.1 | 2.9
  Chronic hepatitis | 26.2 | 22.9
  Vascular lesions | 35.7 | 11.4
  Pathology of biliary obstruction | 4.8 | 5.7
  Lobular hepatitis | 4.8 | 2.9
  Recurrence of initial autoimmune disease | 0.0 | 0.0
  Other | 35.7 | 45.7

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from study start to 28 days after Month 12 or the last dose of study treatment.
Description: All participants who were randomized and received at least one dose of MMF and/or corticosteroids were included in the safety analysis. Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.
Arm/Group | Adjusted MMF + Tacrolimus + CS | Fixed-Dose MMF + Tacrolimus + CS
Serious Adverse Events (participants affected / at risk) | 70/91 | 69/92
Other Adverse Events (participants affected / at risk) | 91/91 | 91/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adjusted MMF + Tacrolimus + CS (N=91) | Fixed-Dose MMF + Tacrolimus + CS (N=92)
Hepatitis C (Infections and infestations) | 3 | 7
Sepsis (Infections and infestations) | 3 | 4
Septic shock (Infections and infestations) | 4 | 1
Peritoneal infection (Infections and infestations) | 2 | 1
Biliary sepsis (Infections and infestations) | 1 | 1
Candida sepsis (Infections and infestations) | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Aspergillosis (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Nocardiosis (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Viral diarrhoea (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Inguinal hernia (Gastrointestinal disorders) | 2 | 4
Ascites (Gastrointestinal disorders) | 2 | 2
Abdominal hernia (Gastrointestinal disorders) | 3 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 2 | 4
Cholangitis (Hepatobiliary disorders) | 2 | 4
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 | 5
Hepatic artery stenosis (Hepatobiliary disorders) | 3 | 2
Biliary fistula (Hepatobiliary disorders) | 3 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 4
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 2
Bile duct necrosis (Hepatobiliary disorders) | 1 | 0
Biliary cyst (Hepatobiliary disorders) | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic artery aneurysm (Hepatobiliary disorders) | 1 | 0
Hepatic ischaemia (Hepatobiliary disorders) | 0 | 1
Hepatic vein stenosis (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 14 | 5
Renal failure (Renal and urinary disorders) | 6 | 6
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 5 | 6
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 4
Graft dysfunction (Injury, poisoning and procedural complications) | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Complications of transplant surgery (Injury, poisoning and procedural complications) | 0 | 1
Complications of transplanted liver (Injury, poisoning and procedural complications) | 1 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1
Multi-organ failure (General disorders) | 5 | 3
General physical health deterioration (General disorders) | 1 | 2
Chest pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 2
Sudden death (General disorders) | 0 | 2
Hyperthermia (General disorders) | 0 | 1
Inflammation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Ulcer haemorrhage (General disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Agranulocytosis (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 2 | 2
Arterial haemorrhage (Vascular disorders) | 1 | 1
Aneurysm (Vascular disorders) | 1 | 0
Angiopathy (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Haemodynamic instability (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Vascular stenosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Cell death (Metabolism and nutrition disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Vocal cord paresis (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 2
Mental disorder (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 3
Cytomegalovirus antibody positive (Investigations) | 0 | 1
Oesophagogastroduodenoscopy (Investigations) | 1 | 0
Biliary anastomosis (Surgical and medical procedures) | 0 | 1
Biliary drainage (Surgical and medical procedures) | 1 | 0
Catheter removal (Surgical and medical procedures) | 0 | 1
Surgical vascular shunt (Surgical and medical procedures) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 0 | 1
Hereditary neuropathic amyloidosis (Congenital, familial and genetic disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Liver transplant rejection (Immune system disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adjusted MMF + Tacrolimus + CS (N=91) | Fixed-Dose MMF + Tacrolimus + CS (N=92)
Diarrhoea (Gastrointestinal disorders) | 31 | 26
Abdominal pain (Gastrointestinal disorders) | 12 | 12
Ascites (Gastrointestinal disorders) | 9 | 11
Constipation (Gastrointestinal disorders) | 8 | 11
Nausea (Gastrointestinal disorders) | 8 | 8
Vomiting (Gastrointestinal disorders) | 10 | 5
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 7
Inguinal hernia (Gastrointestinal disorders) | 2 | 7
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Peritonitis (Gastrointestinal disorders) | 2 | 2
Abdominal hernia (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Coeliac artery stenosis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1
Peritoneal effusion (Gastrointestinal disorders) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Portal venous gas (Gastrointestinal disorders) | 1 | 0
Small bowel angioedema (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 45 | 44
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 13
Neutropenia (Blood and lymphatic system disorders) | 13 | 6
Leukopenia (Blood and lymphatic system disorders) | 14 | 2
Pancytopenia (Blood and lymphatic system disorders) | 11 | 4
Deficiency anaemia (Blood and lymphatic system disorders) | 6 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 3
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 2 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Jaundice acholuric (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Thrombocythaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 13 | 14
Hepatitis C (Infections and infestations) | 7 | 11
Sepsis (Infections and infestations) | 9 | 8
Cytomegalovirus infection (Infections and infestations) | 7 | 6
Staphylococcal infection (Infections and infestations) | 4 | 6
Bronchitis (Infections and infestations) | 2 | 5
Septic shock (Infections and infestations) | 4 | 2
Infection (Infections and infestations) | 4 | 1
Puncture site infection (Infections and infestations) | 3 | 2
Abdominal wall abscess (Infections and infestations) | 2 | 2
Ascites infection (Infections and infestations) | 2 | 2
Enterococcal infection (Infections and infestations) | 4 | 0
Lung infection (Infections and infestations) | 3 | 1
Peritoneal infection (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Oral candidiasis (Infections and infestations) | 0 | 3
Staphylococcal sepsis (Infections and infestations) | 1 | 2
Tonsillitis (Infections and infestations) | 2 | 1
Arthritis bacterial (Infections and infestations) | 1 | 1
Biliary sepsis (Infections and infestations) | 1 | 1
Candida sepsis (Infections and infestations) | 0 | 2
Catheter related infection (Infections and infestations) | 0 | 2
Clostridial infection (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1
Streptococcal infection (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Aspergillosis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1
Citrobacter infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Hepatobiliary infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Infusion site infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Nocardiosis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral fungal infection (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Serratia infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 1 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 15 | 14
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 13
Cell death (Metabolism and nutrition disorders) | 12 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 8
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 5
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Weight fluctuation (Metabolism and nutrition disorders) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypovitaminosis (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 0
Mineral deficiency (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 31 | 31
Venous thrombosis (Vascular disorders) | 7 | 4
Haemodynamic instability (Vascular disorders) | 3 | 7
Haemorrhage (Vascular disorders) | 3 | 4
Hypotension (Vascular disorders) | 3 | 3
Haematoma (Vascular disorders) | 2 | 2
Shock haemorrhagic (Vascular disorders) | 2 | 2
Arterial haemorrhage (Vascular disorders) | 1 | 1
Vein discolouration (Vascular disorders) | 1 | 1
Aneurysm (Vascular disorders) | 1 | 0
Angiopathy (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Phlebitis (Metabolism and nutrition disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Vascular stenosis (Vascular disorders) | 0 | 1
Venous stasis (Vascular disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 24 | 23
Renal failure acute (Renal and urinary disorders) | 22 | 16
Renal impairment (Renal and urinary disorders) | 6 | 8
Oliguria (Renal and urinary disorders) | 4 | 5
Anuria (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 2
Micturition disorder (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1
Renal tubular disorder (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Oedema peripheral (General disorders) | 10 | 17
Pain (General disorders) | 12 | 10
Pyrexia (General disorders) | 11 | 4
Hyperthermia (General disorders) | 8 | 5
Oedema (General disorders) | 7 | 5
Multi-organ failure (General disorders) | 5 | 5
Asthenia (General disorders) | 2 | 6
Inflammation (General disorders) | 2 | 5
Chest pain (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 1 | 2
Hypothermia (General disorders) | 1 | 2
Effusion (General disorders) | 2 | 0
Influenza like illness (General disorders) | 1 | 1
Sudden death (General disorders) | 0 | 2
Catheter site necrosis (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Necrosis (General disorders) | 1 | 0
Polyp (General disorders) | 1 | 0
Ulcer (General disorders) | 1 | 0
Ulcer haemorrhage (General disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 24 | 19
Cholangitis (Hepatobiliary disorders) | 5 | 6
Bile duct stenosis (Hepatobiliary disorders) | 4 | 4
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 | 7
Cytolytic hepatitis (Hepatobiliary disorders) | 4 | 3
Hepatic artery stenosis (Hepatobiliary disorders) | 4 | 3
Jaundice (Hepatobiliary disorders) | 5 | 2
Biliary fistula (Hepatobiliary disorders) | 3 | 3
Portal vein thrombosis (Hepatobiliary disorders) | 5 | 1
Biloma (Hepatobiliary disorders) | 2 | 2
Biliary tract disorder (Hepatobiliary disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2
Biliary cyst (Hepatobiliary disorders) | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Bile duct necrosis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic artery aneurysm (Hepatobiliary disorders) | 1 | 0
Hepatic ischaemia (Hepatobiliary disorders) | 0 | 1
Hepatic vein stenosis (Hepatobiliary disorders) | 0 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 22 | 25
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory gas exchange disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 11 | 14
Insomnia (Psychiatric disorders) | 15 | 10
Agitation (Psychiatric disorders) | 8 | 8
Anxiety (Psychiatric disorders) | 4 | 12
Depression (Psychiatric disorders) | 1 | 6
Delirium (Psychiatric disorders) | 0 | 2
Mental disorder (Psychiatric disorders) | 1 | 1
Affective disorder (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Hallucination, visual (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Headache (Nervous system disorders) | 9 | 10
Tremor (Nervous system disorders) | 8 | 9
Convulsion (Nervous system disorders) | 1 | 4
Febrile convulsion (Nervous system disorders) | 4 | 1
Encephalopathy (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 1 | 2
Dysarthria (Nervous system disorders) | 1 | 2
Epilepsy (Nervous system disorders) | 2 | 1
Paraesthesia (Nervous system disorders) | 1 | 2
Syncope vasovagal (Nervous system disorders) | 3 | 0
Amnesia (Nervous system disorders) | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Polyneuropathy (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 2
Altered state of consciousness (Nervous system disorders) | 1 | 0
Aphonia (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Hyperreflexia (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paresis (Nervous system disorders) | 0 | 1
Psychomotor skills impaired (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Vocal cord paresis (Nervous system disorders) | 0 | 1
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 7 | 6
Seroma (Injury, poisoning and procedural complications) | 4 | 5
Overdose (Injury, poisoning and procedural complications) | 1 | 6
Anastomotic stenosis (Injury, poisoning and procedural complications) | 2 | 4
Eschar (Injury, poisoning and procedural complications) | 3 | 1
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 | 3
Procedural pain (Injury, poisoning and procedural complications) | 4 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 3 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 3 | 0
Graft dysfunction (Injury, poisoning and procedural complications) | 2 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 2 | 0
Complications of transplant surgery (Injury, poisoning and procedural complications) | 0 | 1
Complications of transplanted liver (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Radiation leukopenia (Injury, poisoning and procedural complications) | 1 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Surgical procedure repeated (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Amyotrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Band neutrophil percentage decreased (Investigations) | 4 | 5
Weight decreased (Investigations) | 4 | 5
Red blood cell count decreased (Investigations) | 3 | 4
Liver function test abnormal (Investigations) | 1 | 5
Weight increased (Investigations) | 3 | 2
Gamma-glutamyltransferase increased (Investigations) | 3 | 1
Blood bilirubin increased (Investigations) | 2 | 1
Blood urea increased (Investigations) | 2 | 1
Haematology test abnormal (Investigations) | 0 | 2
Aspiration tracheal (Investigations) | 1 | 0
Blood glucose (Investigations) | 1 | 0
Cytomegalovirus antibody positive (Investigations) | 0 | 1
Oesophagogastroduodenoscopy (Investigations) | 1 | 0
Prothrombin level decreased (Investigations) | 1 | 0
Serum ferritin increased (Investigations) | 0 | 1
Tachycardia (Cardiac disorders) | 6 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 3
Acute coronary syndrome (Cardiac disorders) | 2 | 2
Arrhythmia (Cardiac disorders) | 0 | 3
Bradycardia (Cardiac disorders) | 2 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Pericardial disease (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 3
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Vascular purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 3
Hypersensitivity (Immune system disorders) | 0 | 1
Liver transplant rejection (Immune system disorders) | 0 | 1
Transplant rejection (Immune system disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 2
Visual disturbance (Eye disorders) | 1 | 1
Uveitis (Eye disorders) | 0 | 1
Biliary anastomosis (Surgical and medical procedures) | 0 | 1
Biliary drainage (Surgical and medical procedures) | 1 | 0
Catheter removal (Surgical and medical procedures) | 0 | 1
Skin neoplasm excision (Surgical and medical procedures) | 1 | 0
Surgical vascular shunt (Surgical and medical procedures) | 0 | 1
Hereditary neuropathic amyloidosis (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Alcohol use (Social circumstances) | 0 | 1

LIMITATIONS AND CAVEATS:
Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.